CLINICAL TRIAL: NCT00284999
Title: Soothe Versus Refresh
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pharmaceutical Research Network (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PRN 05-034
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2006-08-22 (Estimated); Status verified 2006-08

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

INTERVENTIONS:
Drug: Soothe
Drug: Refresh Tears

SUMMARY:
To determine the ocular efficacy and safety of Soothe and Refresh Tears.

ELIGIBILITY:
Inclusion Criteria:

* adults with a diagnosis of dry eyes
* Schirmer's with anesthesia grade between 1-7 mm inclusive after five (5) minutes in at least one eye
* a corneal staining grade of greater than or equal to 2 (scale 0-4) in the same qualifying eye as the Schirmer's test

Exclusion Criteria:

* contact lens use during the active treatment periods of the trial
* history of Sjogren's Syndrome
* temporary punctal occlusion that is still effective
* the current or anticipated use during the study of punctual plugs
* current treatment with Restasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33
Dates: Study Completion 2006-08

CONTACTS AND LOCATIONS:
Overall Officials: William C. Stewart, MD, Study Director — Pharmaceutical Research Network, LLC; Penny Asbell, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Christopher Chow, MD, Principal Investigator — Michigan Cornea Associates; Douglas G. Day, MD, Principal Investigator — Coastal Research Associates, LLC
Locations (3):
- United States (3):
  - Coastal Research Associates, LLC, Atlanta, Georgia
  - Michigan Cornea Associates, Southfield, Michigan
  - Mount Sinai School of Medicine, New York, New York